CLINICAL TRIAL: NCT06097091
Title: Effects and Mechanisms of Pain Neuroscience Education on Pain Severity, Disease Severity, Pain Catastrophizing, and Cognitive Function in Patients With Fibromyalgia : A Randomized Controlled Trial
Brief Title: Effects and Mechanisms of Pain Neuroscience Education in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pei-Shan, Tsai, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202305118
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; cognitive function; disease severity; pain catastrophizing; pain neuroscience education; pain severity; quantitative electroencephalography
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: We will employ a triple masking protocol in which the PNE educator, participants, and data collectors will all be blinded to group assignments. In addition, we will mask the group assignment to the data analyzer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Management Education (Active Comparator): Participants in the control group will receive an SME via weekly video calls over 6 weeks.
  Interventions: Other: Self-management education
- Pain Neuroscience Education (Experimental): Participants in the experimental group will receive a 6-week PNE program.
  Interventions: Behavioral: pain neuroscience education

INTERVENTIONS:
Other: Self-management education — A self-management of the FM handbook will be provided. SME will be delivered via weekly video calls over a 6-week period. The video call lasting for 15 minutes, will consist of reviewing the weekly self-management content (5 min), questioning and answering related to the content of the self-management handbook (5 min), and a debriefing session (5 min).
  Arms: Self-Management Education
Behavioral: pain neuroscience education — Participants in the experimental group will receive a 6-week PNE program. The PNE program that is designed to explain pain to the participants will be implemented via 6 individual face-to-face sessions, each lasting for 45 minutes over a 6-week period. Printed take-home materials will be provided to the participants to enhance learning. The goal of PNE is to increase participants' knowledge about pain to help them reconceptualize their beliefs about pain and decrease perceived threats of pain. The content will be composed according to the second edition of the book, "Explain Pain" by Butler and Mosley (2013) as well as etiologies of fibromyalgia. Accordingly, the PI has developed the preliminary PNE content.
  Arms: Pain Neuroscience Education

SUMMARY:
This randomized controlled trials study aims, first, to determine the effectiveness of a nurse-led PNE program designed by a multidisciplinary team, compared with an active control group on pain intensity, fibromyalgia (FM) severity, pain catastrophizing, and cognitive performance in patients with FM. Second, to determine the mediator role of pain catastrophizing in the effects of PNE on outcomes of interest. Third, to explore PNE-induced changes to the brain circuitry using QEEG in patients with FM.

DETAILED DESCRIPTION:
This is a parallel-group, randomized controlled trial (RCT). 98 participants who meet the 2016 American College of Rheumatology diagnostic criteria for FM will be enrolled.

Eligible participants who complete the baseline measurements will be randomly allocated to a PNE group (N = 49) and a self-management education group (N = 49).

Primary outcomes include pain severity determined using the Brief Pain Inventory-Short Form (BPI-SF) and FM severity assessed using the Fibromyalgia Impact Questionnaire-Revised (FIQR).

Secondary outcomes, including pain catastrophizing and sustained attention, will examine using the Pain Catastrophizing Scale (PCS), the Psychomotor Vigilance Test (PVT), and QEEG, respectively.

All outcomes will be measured at 3 different time points: (T0: baseline; T1: immediately after the 6-week intervention period; and T2: 3 months after the intervention period).

Implications:

This will be the first-ever RCT to examine the effectiveness of a Chinese-language PNE program and the first study to determine the brain changes after PNE using QEEG in patients with FM. Once the effectiveness of the PNE and its brain mechanisms are supported by evidence from this trial, it will become a game changer in the management of the FM population. If an evidence-based PNE platform based on the patented training course is subsequently developed, the product will have great potential for commercialization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must read and understand Chinese language.
* According to the 2016 ACR diagnostic criteria, participants' PDS scores more than or equal to 13 points

Exclusion Criteria:

* Subjects who have medical history of traumatic brain injury or neurological disorder.
* Subjects who have present psychopathologic disorder.
* Subjects who are cancer.
* Subjects who are pregnancy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
the Brief Pain Inventory-Short Form (BPI-SF) | baseline; T1 = immediately after PNE; T2 = 3th month after intervention.
  The BPI-SF evaluates pain in different contexts: worst pain, least pain, average pain, and current pain, rated on a 0-10 scale.
the Fibromyalgia Impact Questionnaire Revised (FIQR) | baseline; T1 = immediately after PNE; T2 = 3th month after intervention.
  The FIQR includes 21 questions involving 3 domains: physical function, overall effect of fibromyalgia, and fibromyalgia symptoms (pain, fatigue, unrefreshing sleep, stiffness, anxiety, depression, tenderness to touch, memory, balance, and environmental sensitivity).

SECONDARY OUTCOMES:
Pain Catastrophizing Scale(PCS) | baseline; T1 = immediately after PNE; T2 = 3th month after intervention.
  The PCS is a self-reported questionnaire consisting of 13 items that assess negative emotional and cognitive processes (e.g., helplessness, rumination, pessimism, and magnification of symptoms).
Psychomotor Vigilance Test (PVT) | baseline; T1 = immediately after PNE; T2 = 3th month after intervention.
  The standard 3-minute PVT will be used in this study to assess sustained or vigilant attention. The PVT is performed by recording the response time to visual stimuli, occurring at random inter stimulus intervals.

OTHER OUTCOMES:
Quantitative electroencephalography | baseline; T1 = immediately after PNE; T2 = 3th month after intervention.
  Resting-state EEG measurements with eyes closed will be taken for 10 min using the BrainMaster Discovery 24 EEG device. The participants will be seated with their eyes closed for 20 min before the measurements to achieve this stable/resting state. Five minutes of artifact-free EEG will be used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Shan Tsai, PhD, Study Chair — Taipei Medical University, Taiwan
Locations (1):
- Bio-Behavior Research Laboratory, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No